Study Title:

Patient Education on Labor Analgesia Options

Last updated: 10/31/2018

NCT number: NCT02557555

## Statistical Analysis Plan

In this study, a total of 100 patients received and completed a questionnaire containing 24 questions. For questions involving a Yes/No answer, a test for equality of proportions was utilized to analyze the data. Results were determined to be statistically significant at P < 0.05.